CLINICAL TRIAL: NCT06121375
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2/3 Study to Assess the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Obeticholic Acid Compared to Placebo in Pediatric Subjects With Biliary Atresia, Post-hepatoportoenterostomy
Brief Title: Study to Assess Efficacy, Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Obeticholic Acid (OCA) Compared to Placebo in Pediatric Participants With Biliary Atresia, Post-hepatoportoenterostomy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Intercept made a business decision to terminate the study based on FDA's request for voluntary withdrawal of Ocaliva and the issuance of clinical hold on studies under US IND involving OCA.
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 747-308
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Biliary Atresia
Keywords: Biliary Atresia; Placebo-controlled; Pharmacokinetics; Pharmacodynamics; Obeticholic Acid; Efficacy; Post-hepatoportoenterostomy
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Participants receiving OCA (Active Comparator): Participants will be randomized to receive OCA (starting at 1.5 milligrams [mg] adult equivalent dose [AED]) orally, with water, once daily. Dose will be titrated every 2 weeks in a stepwise manner for the first 6 weeks, starting at 1.5 mg AED and titrating through 3 mg AED to a maximum of 5 mg AED, as tolerated; a discussion with the Medical Monitor is encouraged when determining uptitration if considerable signs or symptoms have arisen. Following the 6-week dose titration phase, participants will continue at the tolerated dose for approximately 24 months in Age Expansion Treatment Phase.
  Interventions: Drug: OCA
- Participants receiving Matching placebo (Placebo Comparator): Participants will be randomized to receive matching placebo orally, with water, once daily. Dose will be titrated every 2 weeks in a stepwise manner for the first 6 weeks, starting at 1.5 mg AED and titrating through 3 mg AED to a maximum of 5 mg AED, as tolerated; a discussion with the Medical Monitor is encouraged when determining uptitration if considerable signs or symptoms have arisen. Following the 6-week dose titration phase, participants will continue at the tolerated dose for approximately 24 months in Age Expansion Treatment Phase.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: OCA — OCA will be administered.
  Arms: Participants receiving OCA
Drug: Matching Placebo — Matching Placebo will be administered.
  Arms: Participants receiving Matching placebo

SUMMARY:
This study will evaluate the efficacy, safety and tolerability, as well as PK/PD of OCA in eligible pediatric participants with biliary atresia with successful hepatoportoenterostomy (HPE, also known as a Kasai portoenterostomy). The double-blind period comprises of 2 phases: dose titration phase and age expansion treatment phase.

ELIGIBILITY:
Inclusion criteria:

* Male or female pediatric participants from birth to <18 years old. Note: Participants aged <2 years old will not be enrolled until after review of safety data during the planned interim analysis and agreement from the Data Safety Monitoring Board (DSMB) that there is sufficient safety data to enroll this age group.
* Diagnosis of non-syndromic biliary atresia.
* Demonstrated successful HPE as defined by total bilirubin <2 milligrams per deciliter (mg/dL) (34.2 micromoles per liter [μmol/L]) at least 3 months post-HPE procedure.

Exclusion criteria:

* Prior liver transplant or active status on transplant list.
* Participants diagnosed with biliary atresia splenic malformation (BASM).
* Conjugated (direct) bilirubin ≥ upper limit of normal (ULN) of site-specific reference range. If conjugated bilirubin is not available: total bilirubin ≥2 mg/dL (34.2 mol/L).
* Platelets <120,000/μL
* International normalized ratio (INR) ≥1.5.
* Current or history of complications of decompensated chronic liver disease including:

  1. Gastroesophageal varices and/or variceal bleeding
  2. Clinically evident ascites related to portal hypertension
  3. Hepatic encephalopathy
  4. Prior placement of portosystemic shunt
  5. Hepatopulmonary syndrome or portopulmonary hypertension
  6. Hepatorenal syndrome
  7. Any evidence of portal hypertension based on imaging (e.g., cavernous transformation of portal vein, abdominal varices, etc.)
  8. Hepatocellular carcinoma
  9. Childs-Pugh B or C
* Height and weight Z-score <-2 per site-specific reference ranges.
* Acholic (pale) stools.
* Aspartate aminotransferase (AST) >4x ULN.
* Alanine aminotransferase >4x ULN
* GGT >500 Units per Liter (U/L)
* On anticoagulation therapy
* Albumin <3.5 grams per deciliter (g/dL).
* Inability to swallow tablets (i.e., tablet or mini-tablet formulations).

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Time to the First Occurrence of Composite Endpoint | Up to Week 64
  To evaluate the effect of OCA compared to placebo in conjunction with established local standard of care on clinical outcomes in participants with biliary atresia who have had a successful Kasai procedure as measured by time to first occurrence of any of the following adjudicated events, derived as composite event endpoint of all-cause death, liver transplant, Pediatric end-stage liver disease (PELD) score ≥17/model of end-stage liver disease (MELD)≥15, Hospitalization (as defined by a stay of 24 hours or greater) for new onset or recurrence of Variceal bleed, hepatic encephalopathy (as defined by a West Haven score of ≥2), Spontaneous bacterial peritonitis (confirmed by diagnostic paracentesis) and Clinically evident ascites related to poral hypertension (diuretic-resistant ascites requiring therapeutic paracentesis at a frequency of at least twice in a month)

SECONDARY OUTCOMES:
Plasma concentration of unconjugated OCA (parent), glyco-OCA, tauro-OCA, and total OCA (molar sum of OCA and its active conjugates) | Up to Week 64
  Plasma concentrations of OCA and its conjugates (glyco-OCA and tauro-OCA) will be determined using validated liquid-chromatography mass spectrometry/mass spectrometry methods
Change from Baseline in Gamma Glutamyl Transferase (GGT) | Baseline and up to Week 64
  Blood samples will be calculated to assess GGT levels.
Change from Baseline in total and direct (conjugated) bilirubin | Baseline and up to Week 64
  Blood samples will be calculated to assess total and direct (conjugated) bilirubin levels.
Change from Baseline in Fibroblast Growth Factor-19 (FGF-19) | Baseline and up to Week 64
  Blood samples will be calculated to assess FGF-19
Change from Baseline in 7-hydroxyl-4-cholesten-3-one (C4) | Baseline and up to Week 64
  Blood samples will be calculated to assess C4
Change from Baseline in endogenous bile acids | Baseline and up to Week 64
  Blood samples will be calculated to assess endogenous bile acids
Change from Baseline in liver stiffness as assessed by transient elastography | Baseline and up to Week 64
Change from Baseline in plasma levels of fat-soluble vitamins (D and K) | Baseline and up to Week 64
  Blood samples will be calculated to assess plasma levels of fat-soluble vitamins (D and K)
Safety and tolerability as assessed by the incidence of treatment-emergent adverse events (TEAEs) including serious adverse events (SAEs) | Up to Week 64

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Szczech, MD, Study Director — Intercept Pharmaceuticals
Locations (24):
- Australia (3):
  - Queensland Childrens Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Childrens Hospital, Parkville, Victoria
- Canada (2):
  - Alberta Childrens Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
- China (5):
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Guangzhou Women And Childrens Medical Center, Guangzhou
  - Children's Hospital of Fudan University, Shanghai
  - Childrens Hospital of Shanghai, Shanghai
  - Children's Hospital of Shanxi, Taiyuan
- Queen Mary Hospital, Hong Kong, Hong Kong
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Shaare-Zedek Medical Center, Jerusalem
- Malaysia (2):
  - Hospital Raja Perempuan Azinab II, Kota Bharu, Kelantan
  - University Malaya Medical Center, Kuala Lumpur
- Starship Child Health, Auckland, New Zealand
- KK Women's and Children's Hospital, Singapore, Singapore
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Chen Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (3):
  - Akdeniz Üniversitesi Tıp Fakültesi Hastanesi Pediatrik Gastroenteroloji, Konyaalti, Antalya
  - Ege Üniversitesi Hastanesi Pediatrik Gastroenteroloji Bölümü, Bornova, İzmir
  - Hacettepe Universitesi ihsan Dogramaci Cocuk Hastansesi, Ankara

IPD SHARING:
Plan to Share IPD: No